CLINICAL TRIAL: NCT04321343
Title: A 36-week, Randomized, Double-blind, Placebo-controlled, Parallel Group Trial to Assess the Efficacy and Safety of PXL065 Versus Placebo in Noncirrhotic Biopsy-proven NonAlcoholic SteatoHepatitis (NASH) Patients
Brief Title: Study of PXL065 in Patients With Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PXL065-003
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Results first posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): PXL065 Dose 1
  Interventions: Drug: PXL065
- Group 2 (Experimental): PXL065 Dose 2
  Interventions: Drug: PXL065
- Group 3 (Experimental): PXL065 Dose 3
  Interventions: Drug: PXL065
- Group 4 (Placebo Comparator): Placebo oral tablet
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: PXL065 — PXL065 oral tablet
  Arms: Group 1; Group 2; Group 3
Drug: Placebo oral tablet — Placebo oral tablet
  Arms: Group 4

SUMMARY:
This study will assess the effect of 3 doses of PXL065 versus placebo on liver fat content in NASH patients after 36 weeks of treatment

DETAILED DESCRIPTION:
The study will be performed in patients with NASH. The primary endpoint will be the assessment of the change in the percentage of liver fat content (assessed by MRI-PDFF).

ELIGIBILITY:
Inclusion Criteria:

* Patients have given written informed consent
* Body mass index (BMI) ≤ 50 kg/m²
* For patients with type 2 diabetes mellitus: either naive of glucose lowering drug or under stable oral glucose lowering drug
* Estimated glomerular filtration rate (eGFR) ≥ 45 mL/min/1.73m²
* Liver fat content ≥ 8% on MRI-PDFF
* Qualifying liver biopsy (NAS) ≥ 4 and fibrosis score F1, F2 or F3
* Effective contraception for women of child bearing potential

Exclusion Criteria:

* Evidence of another form of liver disease
* Evidence of liver cirrhosis
* Evidence of hepatic impairment
* Positive serologic evidence of current infectious liver disease
* History of excessive alcohol intake
* Acute cardiovascular disease within 6 months prior to Randomization
* Any disease which in the Investigator's opinion which in the Investigator's opinion would exclude the patient from the study
* Use of non-permitted concomitant medication
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Study site 11, Chandler, Arizona
  - Study site 12, Glendale, Arizona
  - Study site 13, Tucson, Arizona
  - Study site 21, Tucson, Arizona
  - Study site 17, Chula Vista, California
  - Study site 16, Fresno, California
  - Study site 04, Huntington Park, California
  - Study site 05, Los Angeles, California
  - Study site 22, Orange, California
  - Study site 06, Panorama City, California
  - Study site 07, Santa Ana, California
  - Study site 15, Boca Raton, Florida
  - Study site 31, Fort Myers, Florida
  - Study site 08, Port Orange, Florida
  - Study site 01, Sarasota, Florida
  - Study site 28, West Des Moines, Iowa
  - Study site 18, Kansas City, Kansas
  - Study site 24, Flowood, Mississippi
  - Study site 10, Jackson, Mississippi
  - Study site 27, East Syracuse, New York
  - Study site 14, Fayetteville, North Carolina
  - Study site 29, Summerville, South Carolina
  - Study site 25, Chattanooga, Tennessee
  - Study site 30, Clarksville, Tennessee
  - Study Site 02, Germantown, Tennessee
  - Study site 19, Austin, Texas
  - Study site 09, Edinburg, Texas
  - Study site 23, Edinburg, Texas
  - Pinnacle Clinical Research (Study site 20), San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for the study at 28 sites in the United States between 01Sep2020 and 07Sep2021.
Pre-assignment Details: Following a Screening period of maximum 12 weeks, patients who have met all the applicable Inclusion criteria and none of the Exclusion criteria were to be randomized.
Groups:
- PXL065 7.5 mg QD: PXL065 7.5 mg oral tablet + Placebo oral tablet
- PXL065 15 mg QD: PXL065 15 mg oral tablet + Placebo oral tablet
- PXL065 22.5 mg QD: PXL065 7.5 mg oral tablet + PXL065 15 mg oral tablet
- Placebo: Placebo oral tablets
Period: Overall Study
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Started | 25 | 32 | 30 | 30
Completed the Double-blind Period | 21 | 23 | 27 | 24
Completed | 21 | 23 | 27 | 23
Not Completed | 4 | 9 | 3 | 7
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 6 | 0 | 2
Not completed — Lost to Follow-up | 2 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent to treat set (ITTS), defined as all as-randomized patients who received at least one dose of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo | Total
Number analyzed (Participants) | 25 | 32 | 30 | 30 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 27 | 23 | 23 | 92
  >=65 years | 6 | 5 | 7 | 7 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (17.28) | 54.1 (10.86) | 53.4 (12.36) | 54.8 (10.15) | 53.4 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 14 | 21 | 67
  Male | 11 | 14 | 16 | 9 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 13 | 9 | 41
  Not Hispanic or Latino | 14 | 24 | 17 | 21 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 2
  Asian | 1 | 2 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 22 | 26 | 29 | 29 | 106
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
T2DM status (stratification group) [Count of Participants; unit: Participants]
  T2DM patients | 10 | 13 | 12 | 13 | 48
  Non-T2DM patients | 15 | 19 | 18 | 17 | 69
NASH CRN fibrosis score (stratification group) [Count of Participants; unit: Participants] — This score was determined by a central reader based on stained liver biopsy slide. In the NASH CRN system, fibrosis stage 0 = no fibrosis; stage 1 = centrilobular pericellular fibrosis (or periportal fibrosis in children); stage 2 = centrilobular and periportal fibrosis; stage 3 = bridging fibrosis; and stage 4 = cirrhosis.
  Participants
    F1 | 9 | 11 | 11 | 10 | 41
    F2 or F3 | 16 | 21 | 19 | 20 | 76

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline to Week 36 in the Percentage of Liver Fat Content (LFC) (Assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction [MRI-PDFF])
Description: MRI-PDFF was performed using a standardized imaging protocol, and a central reader analyzed the results. The central reader for this study trained the local imaging centers and provided the imaging manual.
  Relative change from baseline to Week 36 was calculated as follows: (LFC at Week 36 - LFC at baseline) / LFC at baseline x 100.
  The primary analysis was performed for the Intent-to-treat Set (ITTS) using an analysis of covariance (ANCOVA) model adjusting for treatment, for stratification factors, and for the baseline LFC as a continuous covariate. LFC missing values at Week 36 were imputed using a multivariate imputation approach by fully conditional specification regression method assuming Missing At Random Mechanism.
Time Frame: Baseline and Week 36
Population: Intent-to-treat set (ITTS), defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: percentage of change in LFC
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
percentage of change in LFC | -22.900 (7.104) | -18.590 (6.904) | -21.335 (6.446) | 2.413 (6.619)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.0083, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -25.313, 95% CI 2-sided [-44.1036 to -6.5227], Standard Error of Mean 9.587 — Mean difference (final values) is the difference in Least Squares (LS) Means estimated in the ANCOVA model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0237, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -21.003, 95% CI 2-sided [-39.2074 to -2.7991], Standard Error of Mean 9.287 — Mean difference (final values) is the difference in Least Squares (LS) Means estimated in the ANCOVA model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0087, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -23.748, 95% CI 2-sided [-41.4923 to -6.0035], Standard Error of Mean 9.053 — Mean difference (final values) is the difference in Least Squares (LS) Means estimated in the ANCOVA model

2. Primary Outcome: Relative Change From Baseline to Week 36 in the Percentage of LFC (Assessed by MRI-PDFF) (Wilcoxon Test Sensitivity Analysis)
Description: MRI-PDFF was performed using a standardized imaging protocol, and a central reader analyzed the results. The central reader for this study trained the local imaging centers and provided the imaging manual. The sensitivity analysis was performed for the Intent-to-treat Set (ITTS) using a non parametric pairwise Wilcoxon test stratified according to T2DM status and NASH CRN fibrosis scoring system. LFC missing values at Week 36 were imputed using a multivariate imputation approach by fully conditional specification regression method assuming Missing At Random Mechanism.
Time Frame: Baseline and Week 36
Population: Intent-to-treat set (ITTS), defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Median (Inter-Quartile Range); unit: percentage of change in LFC
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
percentage of change in LFC | -26.555 [-42.700 to -5.664] | -25.353 [-36.586 to -9.826] | -24.782 [-48.391 to -9.096] | 0.937 [-21.632 to 26.116]
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.0105, Wilcoxon (Mann-Whitney); Non-parametric pairwaise Wilcoxon tests using a multiple imputation procedure based on the fully conditional specification method; Hodges-Lehmann midpoint estimate = -26.226, 95% CI 2-sided [-46.3208 to -6.1313], Standard Error of Mean 10.252
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0295, Wilcoxon (Mann-Whitney); [statistical method as in outcome 2, analysis 1]; Hodges-Lehmann midpoint estimate = -21.496, 95% CI 2-sided [-40.8475 to -2.1451], Standard Error of Mean 9.873
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0127, Wilcoxon (Mann-Whitney); [statistical method as in outcome 2, analysis 1]; Hodges-Lehmann midpoint estimate = -24.290, 95% CI 2-sided [-43.3920 to -5.1884], Standard Error of Mean 9.746

3. Secondary Outcome: Absolute Change From Baseline to Week 36 in the Percentage of LFC (Assessed by MRI-PDFF)
Description: MRI-PDFF was performed using a standardized imaging protocol, and a central reader analyzed the results. The central reader for this study trained the local imaging centers and provided the imaging manual.
  Absolute change from baseline to Week 36 was calculated as follows: LFC at Week 36 - LFC at baseline.
  The analysis of the absolute change in LFC was performed for the Intent-to-treat Set (ITTS) using an ANCOVA model adjusting for treatment, for stratification factors, and for the baseline LFC as a continuous covariate. LFC missing values at Week 36 were imputed using a multivariate imputation approach by fully conditional specification regression method assuming Missing At Random Mechanism.
Time Frame: Baseline and Week 36
Population: Intent-to-treat set (ITTS), defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: percentage of LFC
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
percentage of LFC | -4.934 (1.381) | -4.360 (1.305) | -4.584 (1.207) | -0.263 (1.228)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.0105, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -4.671, 95% CI 2-sided [-8.2463 to -1.0957], Standard Error of Mean 1.824 — Mean difference (final values) is the difference in Least Squares (LS) Means estimated in the ANCOVA model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0188, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -4.097, 95% CI 2-sided [-7.5140 to -0.6799], Standard Error of Mean 1.743 — Mean difference (final values) is the difference in Least Squares (LS) Means estimated in the ANCOVA model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0105, ANCOVA; ANCOVA model using a multiple imputation procedure based on the fully conditional specification method; Mean Difference (Final Values) = -4.321, 95% CI 2-sided [-7.6307 to -1.0104], Standard Error of Mean 1.689 — Mean difference (final values) is the difference in Least Squares (LS) Means estimated in the ANCOVA model

4. Secondary Outcome: Percentage of Responders (Relative Reduction of at Least 30% in LFC) at Week 36
Description: Responders were defined as patients who achieved a clinically meaningful relative reduction of at least 30% in LFC from baseline to Week 36 as assessed by MRI-PDFF
Time Frame: Baseline and Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
  For patients with missing Week 36/Early termination, multiple imputation by fully conditional specification methods was used for analysis, although the n counts and percentages reflect only the observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 20 | 24 | 27 | 25
Participants
  Responder | 8 | 11 | 12 | 5
  Non-responder | 12 | 13 | 15 | 20
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.1634, Cochran-Mantel-Haenszel; CMH with multiple imputation; Odds Ratio (OR) = 2.61, 95% CI 2-sided [0.677 to 10.087]
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0722, Cochran-Mantel-Haenszel; CMH with multiple imputation; Odds Ratio (OR) = 3.26, 95% CI 2-sided [0.899 to 11.831]
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0703, Cochran-Mantel-Haenszel; CMH with multiple imputation; Odds Ratio (OR) = 3.17, 95% CI 2-sided [0.909 to 11.052]

5. Secondary Outcome: Change From Baseline to Week 36 in Alanine Amino Transferase (ALT)
Description: Blood samples were collected, handled and stored according to the instructions described in the laboratory manual and all measurements were performed at a central laboratory.
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
U/L | -18.4 (6.0) | -13.6 (5.9) | -6.7 (5.4) | -11.9 (5.6)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.4318, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -6.5, 95% CI 2-sided [-22.66 to 9.72], Standard Error of Mean 8.2 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.8382, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-17.37 to 14.10], Standard Error of Mean 8.0 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.4982, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 5.2, 95% CI 2-sided [-9.92 to 20.33], Standard Error of Mean 7.7 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

6. Secondary Outcome: Percentage of Responders (Normalization of ALT)
Description: Normalization of ALT was analyzed in the subset of patients with baseline greater than the upper reference range. Patients were classed as responders if ALT normalized, i.e. decreased to < upper reference range at a post baseline visit.
Time Frame: Baseline to Week 36
Population: Subset of patients with increased baseline value from the ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 17 | 24 | 24 | 18
Participants
  Responder | 3 | 12 | 10 | 4
  Non-responder | 14 | 12 | 14 | 14
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.7137, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.131 to 3.935]
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0597, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.70, 95% CI 2-sided [0.937 to 14.580]
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.1749, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.61, 95% CI 2-sided [0.655 to 10.430]

7. Secondary Outcome: Change From Baseline to Week 36 in Aspartate Amino Transferase (AST)
Description: as for outcome 5
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
U/L | -10.1 (6.5) | -10.2 (6.3) | -4.9 (5.8) | -7.2 (6.0)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.7449, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-20.15 to 14.43], Standard Error of Mean 8.8 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.7255, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-19.93 to 13.90], Standard Error of Mean 8.6 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.7755, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-13.89 to 18.59], Standard Error of Mean 8.2 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

8. Secondary Outcome: Percentage of Responders (Normalization of AST)
Description: Normalization of AST was analyzed in the subset of patients with baseline greater than the upper reference range. Patients were classed as responders if AST normalized, i.e. decreased to < upper reference range at a post baseline visit.
Time Frame: Baseline to Week 36
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 17 | 17 | 19 | 16
Participants
  Responder | 9 | 4 | 11 | 4
  Non-responder | 8 | 13 | 8 | 12
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.1325, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.12, 95% CI 2-sided [0.703 to 13.806]
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.9918, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.201 to 4.898]
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0410, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.78, 95% CI 2-sided [1.053 to 21.714]

9. Secondary Outcome: Change From Baseline to Week 36 in Gamma Glutamyltransferase (GGT)
Description: as for outcome 5
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
U/L | -12.2 (7.6) | -21.8 (7.5) | -6.9 (6.9) | -4.2 (7.1)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.4413, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -7.9, 95% CI 2-sided [-28.25 to 12.36], Standard Error of Mean 10.3 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0859, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -17.6, 95% CI 2-sided [-37.63 to 2.50], Standard Error of Mean 10.2 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.7887, Mixed Models Analysis; Mixed Model Repeated Measures; Median Difference (Final Values) = -2.7, 95% CI 2-sided [-22.31 to 16.97], Standard Error of Mean 10.0 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

10. Secondary Outcome: Change From Baseline to Week 36 in Alkaline Phosphatase (ALP)
Description: as for outcome 5
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
U/L | -2.8 (2.7) | -8.0 (2.7) | -5.8 (2.5) | 3.1 (2.6)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.1166, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-13.19 to 1.47], Standard Error of Mean 3.7 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0030, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -11.0, 95% CI 2-sided [-18.26 to -3.80], Standard Error of Mean 3.7 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0131, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -8.8, 95% CI 2-sided [-15.79 to -1.87], Standard Error of Mean 3.5 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

11. Secondary Outcome: Change From Baseline to Week 36 in Pro-C3
Description: Pro-C3 is the released N-terminal pro-peptide of type III collagen. It is a fibrosis marker.
  Blood samples were collected, handled and stored according to the instructions described in the laboratory manual and all measurements were performed at a central laboratory.
Time Frame: Baseline and Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
ng/mL | -2.054 (1.182) | -1.753 (1.089) | -2.481 (1.050) | -1.041 (0.893)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.4963, Regression, Linear; Mean Difference (Final Values) = -1.013, 95% CI 2-sided [-3.9701 to 1.9436], Standard Error of Mean 1.481 — Mean difference (final values) is the difference in LS Means estimated in the linear regression
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.6131, Regression, Linear; Mean Difference (Final Values) = -0.712, 95% CI 2-sided [-3.5109 to 2.0866], Standard Error of Mean 1.402 — Mean difference (final values) is the difference in LS Means estimated in the linear regression
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.2939, Regression, Linear; Mean Difference (Final Values) = -1.441, 95% CI 2-sided [-4.1593 to 1.2779], Standard Error of Mean 1.362 — Mean difference (final values) is the difference in LS Means estimated in the linear regression

12. Secondary Outcome: Change From Baseline to Week 36 in Enhanced Liver Fibrosis (ELF) Score
Description: ELF score is an extracellular matrix marker set consisting of tissue inhibitor of metalloproteinases 1 (TIMP-1), amino-terminal propeptide of type III procollagen (PIIINP) and hyaluronic acid (HA) showing good correlations with fibrosis stages in chronic liver disease.The set cutoffs for this scoring are: ELF < 7.7: no to mild fibrosis; ELF between 7.7 - 9.8: moderate fibrosis; ELF between 9.8 - 11.3: severe fibrosis; and ELF > or = 11.3: cirrhosis.
  Blood samples used for TIMP-1, PIIINP and HA were collected, handled and stored according to the instructions described in the laboratory manual and all measurements were performed at a central laboratory.
Time Frame: Baseline and Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
Score | -0.142 (0.168) | -0.206 (0.153) | -0.358 (0.130) | -0.079 (0.130)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.7672, Regression, Linear; Mean Difference (Final Values) = -0.063, 95% CI 2-sided [-0.4845 to 0.3589], Standard Error of Mean 0.211 — Mean difference (final values) is the difference in LS Means estimated in the linear regression
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.5233, Regression, Linear; Mean Difference (Final Values) = -0.127, 95% CI 2-sided [-0.5216 to 0.2678], Standard Error of Mean 0.198 — Mean difference (final values) is the difference in LS Means estimated in the linear regression
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.1263, Regression, Linear; Mean Difference (Final Values) = -0.279, 95% CI 2-sided [-0.6376 to 0.0805], Standard Error of Mean 0.180 — Mean difference (final values) is the difference in LS Means estimated in the linear regression

13. Secondary Outcome: Change From Baseline to Week 36 in Fibrosis-4 (Fib-4) Score
Description: Fib-4 score is a non invasive method based on clinical determinations that indicates the level of fibrosis/ scarring of the liver. The set cutoffs for this scoring are: Fib-4 < 1.45: absence of cirrhosis; Fib-4 between 1.45 - 3.25: inconclusive and Fib-4 > 3.25: cirrhosis.
  Fib-4 score was calculated as (Age [years] × AST [U/L]) / (platelet [10^9/L] × √[ALT [U/L]]). Blood samples used for AST, ALT and platelet counts were collected, handled and stored according to the instructions described in the laboratory manual and all measurements were performed at a central laboratory.
Time Frame: Baseline and Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
Score | -0.040 (0.127) | -0.107 (0.124) | -0.198 (0.109) | -0.012 (0.110)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.8662, Regression, Linear; Mean Difference (Final Values) = -0.028, 95% CI 2-sided [-0.3559 to 0.3002], Standard Error of Mean 0.165 — Mean difference (final values) is the difference in LS Means estimated in the linear regression
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.5726, Regression, Linear; Mean Difference (Final Values) = -0.094, 95% CI 2-sided [-0.4253 to 0.2369], Standard Error of Mean 0.166 — Mean difference (final values) is the difference in LS Means estimated in the linear regression
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.2289, Regression, Linear; Mean Difference (Final Values) = -0.186, 95% CI 2-sided [-0.4907 to 0.1192], Standard Error of Mean 0.153 — Mean difference (final values) is the difference in LS Means estimated in the linear regression

14. Secondary Outcome: Change From Baseline to Week 36 in NAFLD Fibrosis Score
Description: The NFS is based on a combination of clinical and laboratory measurements (i.e. age, glycemia, BMI, platelet, albumin and AST/ALT ratio). The set cutoffs for this scoring are: < -1.455 for exclusion of advance fibrosis, > -1.455 to < or = 0.675 for indetermined, and > 0.675 for presence of advance fibrosis.
  NFS was calculated as: 1.675 + 0.037 x age (years) + 0.094 x BMI (kg/m²) + 1.13 x Impaired Fasting Glucose or Diabetes (yes =1; no=0) + 0.99 x AST/ALT ratio - 0.013 x platelet (10^9/L) - 0.66 x albumin (g/dL)
Time Frame: Baseline and Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
Score | 0.170 (0.192) | -0.006 (0.188) | -0.264 (0.167) | 0.215 (0.167)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.8595, Regression, Linear; Mean Difference (Final Values) = -0.045, 95% CI 2-sided [-0.5509 to 0.4607], Standard Error of Mean 0.254 — Mean difference (final values) is the difference in LS Means estimated in the linear regression
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.3776, Regression, Linear; Mean Difference (Final Values) = -0.222, 95% CI 2-sided [-0.7194 to 0.2759], Standard Error of Mean 0.250 — Mean difference (final values) is the difference in LS Means estimated in the linear regression
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0424, Regression, Linear; Mean Difference (Final Values) = -0.480, 95% CI 2-sided [-0.9426 to 0.0170], Standard Error of Mean 0.232 — Mean difference (final values) is the difference in LS Means estimated in the linear regression

15. Secondary Outcome: Improvement of at Least 1 Point in NASH CRN Fibrosis Score From Baseline to Week 36
Description: Improvement in fibrosis is defined as a decrease of at least one stage in NASH CRN fibrosis score.
Time Frame: Baseline and Week 36
Population: Patients With Week 36 Assessment from the Intent-to-treat set (ITTS), defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 21 | 22 | 26 | 23
Participants
  Responder | 9 | 11 | 9 | 4
  Non-responder | 12 | 11 | 17 | 19
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.1084, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.31, 95% CI 2-sided [0.775 to 14.152]
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0562, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.11, 95% CI 2-sided [0.959 to 17.594]
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.3333, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.87, 95% CI 2-sided [0.501 to 6.948]

16. Secondary Outcome: Improvement in NAS of at Least 2 Points With no Worsening in NASH CRN Fibrosis Score From Baseline to Week 36
Description: NAS is the NAFLD activity score, calculated as the sum of steatosis, lobular inflammation and ballooning scores. Improvement in NAS is defined as a decrease of at least 2 points. No worsening in NASH CRN fibrosis score means that the score remained stable or decreased.
Time Frame: Baseline and Week 36
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 21 | 22 | 26 | 23
Participants
  Responder | 8 | 11 | 13 | 7
  Non-responder | 13 | 11 | 13 | 16
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.7677, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.345 to 4.230]
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.4828, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.434 to 6.012]
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.2711, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.598 to 6.486]

17. Secondary Outcome: NASH Resolution With no Worsening in NASH CRN Fibrosis Score at Week 36
Description: NASH resolution is defined as a NAS score of 0-1 for inflammation, 0 for ballooning, and any value for steatosis. No worsening in NASH CRN fibrosis score means that the score remained stable or decreased.
Time Frame: Baseline and Week 36
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 21 | 22 | 26 | 23
Participants
  Responder | 8 | 8 | 8 | 7
  Non-responder | 13 | 14 | 18 | 16
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.5981, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.376 to 5.547]
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.6228, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.363 to 5.572]
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.8799, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.245 to 3.323]

18. Secondary Outcome: NASH Resolution With Improvement of at Least 1 Point in NASH CRN Fibrosis Score at Week 36
Description: NASH resolution is defined as a NAS score of 0-1 for inflammation, 0 for ballooning, and any value for steatosis. Improvement in fibrosis is defined as a decrease of at least one stage in NASH CRN fibrosis score.
Time Frame: Baseline and Week 36
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 21 | 22 | 26 | 23
Participants
  Responder | 7 | 7 | 4 | 3
  Non-responder | 14 | 15 | 22 | 20
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.1474, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.28, 95% CI 2-sided [0.625 to 17.208]
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.2620, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.65, 95% CI 2-sided [0.481 to 14.631]
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.6935, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.117 to 4.133]

19. Secondary Outcome: Change From Baseline to Week 36 in Glycated Hemoglobin (HbA1c)
Description: as for outcome 5
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
percentage of glycated hemoglobin | 0.14 (0.11) | -0.06 (0.10) | -0.20 (0.10) | 0.21 (0.10)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.6384, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.350 to 0.215], Standard Error of Mean 0.14 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0549, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.547 to 0.006], Standard Error of Mean 0.14 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0030, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.683 to -0.142], Standard Error of Mean 0.14 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

20. Secondary Outcome: Change From Baseline to Week 36 in Fasting Plasma Glucose (FPG)
Description: as for outcome 5
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
mmol/L | 0.147 (0.286) | 0.361 (0.278) | 0.205 (0.251) | 0.198 (0.269)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.8961, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.051, 95% CI 2-sided [-0.8165 to 0.7149], Standard Error of Mean 0.389 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.6710, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.163, 95% CI 2-sided [-0.5935 to 0.9204], Standard Error of Mean 0.384 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.9846, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.007, 95% CI 2-sided [-0.7092 to 0.7233], Standard Error of Mean 0.364 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

21. Secondary Outcome: Change From Baseline to Week 36 in Serum Insulin
Description: as for outcome 5
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
pmol/L | -78.08 (28.01) | -39.76 (26.71) | -56.55 (23.40) | 6.85 (24.06)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.0216, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -84.93, 95% CI 2-sided [-157.306 to -12.558], Standard Error of Mean 36.75 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.1931, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -46.61, 95% CI 2-sided [-116.957 to 23.738], Standard Error of Mean 35.72 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0581, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -63.40, 95% CI 2-sided [-129.002 to 2.194], Standard Error of Mean 33.31 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

22. Secondary Outcome: Change From Baseline to Week 36 in Serum C-peptide
Description: as for outcome 5
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
nmol/L | -0.205 (0.116) | -0.222 (0.110) | -0.250 (0.095) | 0.051 (0.102)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.0958, Mixed Models Analysis; Mixed Models Analysis; Mean Difference (Final Values) = -0.256, 95% CI 2-sided [-0.5577 to 0.0456], Standard Error of Mean 0.153 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0659, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.273, 95% CI 2-sided [-0.5648 to 0.0181], Standard Error of Mean 0.148 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0297, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.301, 95% CI 2-sided [-0.5728 to -0.0300], Standard Error of Mean 0.138 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

23. Secondary Outcome: Change From Baseline to Week 36 in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: HOMA-IR was calculated as: Serum C-peptide (ng/mL) × FPG (mg/dL) / 405 Blood samples were collected, handled and stored according to the instructions described in the laboratory manual and all measurements were performed at a central laboratory.
  HOMA-IR is an indicator of insulin resistance. The higher the value, the greater the insulin resistance. There is no minimum or maximum index score.
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Index
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
Index | -0.086 (0.134) | -0.123 (0.127) | -0.210 (0.106) | 0.111 (0.116)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.2606, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.197, 95% CI 2-sided [-0.5423 to 0.1476], Standard Error of Mean 0.175 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.1709, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.234, 95% CI 2-sided [-0.5690 to 0.1016], Standard Error of Mean 0.170 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0400, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.321, 95% CI 2-sided [-0.6274 to -0.0148], Standard Error of Mean 0.155 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

24. Secondary Outcome: Change From Baseline to Week 36 in Quantitative Insulin Sensitivity Check Index (QUICKI)
Description: The QUICKI was calculated as: 1 / (log (FPG [mg/dL]) + log (C-peptide [ng/mL])).
  Blood samples were collected, handled and stored according to the instructions described in the laboratory manual and all measurements were performed at a central laboratory.
  QUICKI is an indicator of insulin resistance. Lower numbers reflect greater insulin resistance. There is no minimum or maximum index score.
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Index
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
Index | 0.006 (0.009) | 0.007 (0.009) | 0.012 (0.008) | -0.005 (0.008)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.3955, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.011, 95% CI 2-sided [-0.0139 to 0.0351], Standard Error of Mean 0.012 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.3081, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.012, 95% CI 2-sided [-0.0115 to 0.0362], Standard Error of Mean 0.012 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.1374, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.0053 to 0.0383], Standard Error of Mean 0.011 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

25. Secondary Outcome: Change From Baseline to Week 36 in Adipo-IR
Description: The Adipo-IR was calculated as: Fasting serum Free Fatty Acids (mmol/L) x Fasting serum insulin (μIU/mL) Blood samples were collected, handled and stored according to the instructions described in the laboratory manual and all measurements were performed at a central laboratory.
  The Adipo-IR is a marker of adipose tissue insulin resistance. Higher the value, the greater the insulin resistance. There is no minimum or maximum index score.
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Index
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
Index | -36.18 (16.53) | -17.01 (13.78) | -41.87 (12.37) | 12.77 (13.03)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.0199, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -48.94, 95% CI 2-sided [-90.073 to -7.817], Standard Error of Mean 20.86 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.1120, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -29.77, 95% CI 2-sided [-66.558 to 7.009], Standard Error of Mean 18.66 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0026, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = -54.64, 95% CI 2-sided [-89.935 to -19.340], Standard Error of Mean 17.90 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

26. Secondary Outcome: Change From Baseline to Week 36 in Adiponectin
Description: as for outcome 5
Time Frame: Baseline to Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: µg/mL
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
µg/mL | 1.532 (0.679) | 2.688 (0.646) | 4.734 (0.624) | -0.143 (0.595)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.0639, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 1.674, 95% CI 2-sided [-0.0980 to 3.4470], Standard Error of Mean 0.896 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0014, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 2.831, 95% CI 2-sided [1.1149 to 4.5464], Standard Error of Mean 0.867 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 4.876, 95% CI 2-sided [3.1982 to 6.5543], Standard Error of Mean 0.848 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

27. Secondary Outcome: Change From Baseline to Week 36 in Weight
Description: Body weight was measured using a scale with appropriate resolution, placed on a stable, flat surface. Shoes, bulky layers of clothing, and jackets had to be removed so that only light clothing remained.
Time Frame: Baseline to Week 36
Population: Safety Set, defined as all as-treated patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
kg | 1.080 (0.673) | 2.356 (0.636) | 0.577 (0.603) | -0.103 (0.623)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.1944, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 1.183, 95% CI 2-sided [-0.6080 to 2.9748], Standard Error of Mean 0.909 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0056, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 2.459, 95% CI 2-sided [0.7268 to 4.1907], Standard Error of Mean 0.879 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.4288, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.680, 95% CI 2-sided [-1.0111 to 2.3720], Standard Error of Mean 0.858 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

28. Post Hoc Outcome: Change From Baseline to Week 36 in PIIINP
Description: PIIINP is the amino-terminal propeptide of type III procollagen. It is a fibrosis marker.
  Blood samples were collected, handled and stored according to the instructions described in the laboratory manual and all measurements were performed at a central laboratory.
Time Frame: Baseline and Week 36
Population: ITTS, defined as all as-randomized patients who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: µg/mL
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
µg/mL | -2.385 (0.875) | -2.732 (0.796) | -3.354 (0.674) | -1.134 (0.672)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.2564, Regression, Linear; Mean Difference (Final Values) = -1.251, 95% CI 2-sided [-3.4307 to 0.9295], Standard Error of Mean 1.093 — Mean difference (final values) is the difference in LS Means estimated in the linear regression
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.1222, Regression, Linear; Mean Difference (Final Values) = -1.598, 95% CI 2-sided [-3.6348 to 0.4392], Standard Error of Mean 1.021 — Mean difference (final values) is the difference in LS Means estimated in the linear regression
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0206, Regression, Linear; Mean Difference (Final Values) = -2.220, 95% CI 2-sided [-4.0880 to -0.3510], Standard Error of Mean 0.936 — Mean difference (final values) is the difference in LS Means estimated in the linear regression

29. Post Hoc Outcome: Improvement of at Least 2 Points in NAS
Description: NAS is the NAFLD activity score, calculated as the sum of steatosis, lobular inflammation and ballooning scores. Improvement in NAS is defined as a decrease of at least 2 points.
Time Frame: Baseline and Week 36
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 21 | 22 | 26 | 23
Participants
  Responder | 9 | 11 | 15 | 7
  Non-responder | 12 | 11 | 11 | 16
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.5221, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.436 to 5.201]
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.4828, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.434 to 6.012]
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.0914, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.87, 95% CI 2-sided [0.853 to 9.636]

30. Post Hoc Outcome: Improvement of at Least 1 Point in NASH CRN Fibrosis Score With no Worsening of NASH From Baseline to Week 36
Description: Improvement in fibrosis is defined as a decrease of at least one stage in NASH CRN fibrosis score. No worsening of NASH is defined as no increase in steatosis, inflammation or ballooning
Time Frame: Baseline and Week 36
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 21 | 22 | 26 | 23
Participants
  Responder | 8 | 11 | 8 | 4
  Non-responder | 13 | 11 | 18 | 19
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.1854, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.71, 95% CI 2-sided [0.628 to 11.679]
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0562, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.11, 95% CI 2-sided [0.959 to 17.594]
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.5223, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.398 to 5.880]

31. Post Hoc Outcome: Change in Weight Excluding Week 36 for One Patient (Erroneous Data), and Excluding Patients With Weight Loss > 10kg From Baseline to Week 36
Description: as for outcome 27
Time Frame: Baseline to Week 36
Population: Safety Set, defined as all as-treated patients who received at least one dose of study treatment, Excluding Week 36 for one patient (erroneous data), and Excluding Patients With Weight Loss > 10kg from Baseline to Week 36.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
Number analyzed (Participants) | 25 | 32 | 30 | 30
kg | 0.599 (0.656) | 2.304 (0.614) | 0.543 (0.583) | 0.319 (0.612)
Statistical Analysis 1: Comparison: PXL065 7.5 mg QD vs Placebo; Test type: Superiority; p = 0.7532, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.280, 95% CI 2-sided [-1.4749 to 2.0356], Standard Error of Mean 0.891 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 2: Comparison: PXL065 15 mg QD vs Placebo; Test type: Superiority; p = 0.0216, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 1.985, 95% CI 2-sided [0.2946 to 3.6763], Standard Error of Mean 0.858 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model
Statistical Analysis 3: Comparison: PXL065 22.5 mg QD vs Placebo; Test type: Superiority; p = 0.7893, Mixed Models Analysis; Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.224, 95% CI 2-sided [-1.4283 to 1.8771], Standard Error of Mean 0.838 — Mean difference (final values) is the difference in LS Means estimated in the MMRM model

ADVERSE EVENTS:
Time Frame: All AEs were collected from the time of ICF signature to the End-of-study Visit, ie 38 weeks on average.
Description: Only events that occur after the first dose intake of IMP of the Double-blind (DB) treatment period or if they were present prior to the first intake of IMP of the DB treatment period and increased in severity or relationship to IMP after the first intake of IMP of the DB treatment period were considered as Treatment Emergent Adverse Events (TEAEs).
  Only TEAEs (regardless of the relationship) are presented in this section.
Arm/Group | PXL065 7.5 mg QD | PXL065 15 mg QD | PXL065 22.5 mg QD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/32 | 0/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 1/25 | 3/32 | 1/30 | 2/30
Other Adverse Events (participants affected / at risk) | 15/25 | 19/32 | 19/30 | 14/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PXL065 7.5 mg QD (N=25) | PXL065 15 mg QD (N=32) | PXL065 22.5 mg QD (N=30) | Placebo (N=30)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PXL065 7.5 mg QD (N=25) | PXL065 15 mg QD (N=32) | PXL065 22.5 mg QD (N=30) | Placebo (N=30)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 7 (7) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (5) | 2 (2) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (4) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (7) | 8 (12) | 7 (9) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 3 (4) | 3 (3)
Fatigue (General disorders) | 4 (4) | 0 (0) | 1 (1) | 3 (5)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 4 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 4 (5) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of this trial included a relatively small sample size and treatment duration. However, given a close relationship to the parent molecule, pioglitazone, the potential for unforeseen safety issues is low and the present results can be viewed as confirmatory with respect to efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT04321343/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT04321343/SAP_001.pdf